CLINICAL TRIAL: NCT07177885
Title: Tryptophan as a Modulating Factor in the Antimigraine Efficacy of Triptans
Acronym: TRP-Triptans
Status: Not yet recruiting | Type: Observational
Sponsor: University Hospital, Clermont-Ferrand (Other)
Collaborators: University of the Basque Country (UPV/EHU) (Other); Lariboisière Hospital (Unknown)
Responsible Party: Sponsor
Other Study IDs: RBHP 2025 MOISSET 4; 2025-A01152-47 (Other: 2025-A01152-47)
Record Dates: First submitted 2025-09-10; First posted 2025-09-17 (Actual); Last update posted 2025-09-24 (Actual); Status verified 2025-09

CONDITIONS: Migraine
Keywords: Triptan; Tryptophan; inflammatory diseases
MeSH Terms: conditions — Migraine Disorders | interventions — Blood Specimen Collection

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples Without DNA — Blood
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Migraineurs responding to triptans: Blood collection
  Interventions: Biological: Blood collection
- Migraine sufferers resistant to triptans: Blood collection
  Interventions: Biological: Blood collection

INTERVENTIONS:
Biological: Blood collection — Blood sampling. For patients who have had their cerebrospinal fluid sample taken as part of their treatment, a surplus sample will be used to perform the same measurements.

SUMMARY:
Migraine is a leading cause of disability, and while triptans are commonly used to treat migraine attacks, over 20% of patients don't respond well to them. This study aims to understand why some people don't benefit from triptans. One key focus is tryptophan, an amino acid that plays a role in migraine and is involved in producing serotonin, which affects pain and inflammation. The study will compare levels of tryptophan and its by-products in patients who respond well to triptans versus those who don't. It will also look at how conditions like inflammatory bowel disease may affect tryptophan absorption. The goal is to improve migraine treatments tailored to different patient needs, though participants may not experience immediate personal benefits.

DETAILED DESCRIPTION:
Migraine is a leading cause of disability worldwide. Triptans are medications used to treat migraine attacks. They work mainly in two ways: by narrowing the blood vessels in the brain and by stopping the release of substances that cause pain and inflammation. Triptans help relieve migraine pain and other symptoms, like digestive problems, light sensitivity, and disability during an attack. However, more than 20% of patients do not respond well to these medications, and the reasons for this are not well understood.

Tryptophan is an essential amino acid, which means it must come from food because the body cannot produce it. Tryptophan plays an important role in migraines, especially through its by-products, such as serotonin and kynurenine. Research has shown that problems with tryptophan metabolism can make migraines worse, along with other sensory symptoms.

Although no study has directly linked tryptophan to the effectiveness of triptans, the investigators found in a preclinical study that a low-tryptophan diet could reduce the effectiveness of sumatriptan, one of the most commonly used triptans. A deficiency in tryptophan can occur when the body has trouble absorbing it from the intestines. Conditions like inflammatory bowel diseases (such as irritable bowel syndrome or Crohn's disease) or diabetes can affect this absorption, which might reduce the body's ability to process tryptophan.

This study aims to better understand how tryptophan might affect resistance to triptans in migraine patients. The investigators will compare blood levels of tryptophan and its by-products in patients who respond well to triptans versus those who do not. If participants are having a lumbar puncture as part of their regular check-up, the investigators will also examine these substances in the cerebrospinal fluid. Additionally, the investigators will explore any connection between tryptophan metabolism and inflammatory bowel disease.

ELIGIBILITY:
Inclusion Criteria:

* Cisgender women, premenopausal, aged 18 to 50 years.
* Cisgender men, aged 18 to 50 years.
* Diagnosed with migraine (according to ICHD-3 criteria).
* Diagnosed as responders or non-responders to triptans (according to the criteria of Sacco et al., 2022).
* Permitted comparison groups include: triptans used alone or in combination with other migraine treatments (e.g., NSAIDs, acetaminophen, ergotamine, opioids, antiemetics).
* All routes of administration and all dosages.
* Affiliation with a social security system.

Exclusion Criteria:

* Patients under guardianship, curatorship, deprivation of liberty, or legal protection
* Pregnant and breastfeeding women

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — * Cisgender women, premenopausal, between 18 and 50 years old.
  * Cisgender men between 18 and 50 years old.
Study Population: Participants in the study will be recruited from the following centers:
  * Centre 01: CHU de Clermont-Ferrand, Gabriel Montpied site, located at 58 Rue Montalembert, 63000 Clermont-Ferrand, France.
  * Centre 02: Headache Emergency Center, Hôpital Lariboisière, located at 2 Rue Ambroise Paré, 75010 Paris, France.
Sampling Method: Probability Sample
Enrollment: 144 (Estimated)
Dates: Start 2025-11 (Estimated); Primary Completion 2027-11 (Estimated); Study Completion 2028-11 (Estimated)

PRIMARY OUTCOMES:
Plasma tryptophan levels | Baseline
  Variation in plasma tryptophan levels between triptan-resistant and triptan-responsive migraine patients.

SECONDARY OUTCOMES:
Serotonin levels | Baseline
  Variation in plasma serotonin levels between triptan-resistant and triptan-responsive migraine patients.
Kynurenine levels | Baseline
  Variation in plasma kynurenine levels between triptan-resistant and triptan-responsive migraine patients.
Levels of neutral amino acids | Baseline
  Variation in plasma levels of neutral amino acids between triptan-resistant and triptan-responsive migraine patients.
Levels of cytokines (IL-6, IL-10, IL-1α, IL-1β) | Baseline
  Variation in plasma levels of cytokines (IL-6, IL-10, IL-1α, IL-1β) between triptan-resistant and triptan-responsive migraine patients.
Dietary tryptophan intake | Baseline
  Dietary tryptophan intake via a self-questionnaire on eating habits
Inflammatory bowel disorders | Baseline
  Presence/absence of inflammatory bowel disorders
Blood nutritional biomarkers | Baseline
  Variation in blood nutritional biomarkers (glycemia, cholesterol)

OTHER OUTCOMES:
Hospital Anxiety and Depression Scale | Baseline
  Tool for assessing levels of anxiety and depression in patients
Headache Impact | Baseline
  The HIT-6 will be used to assess the impact of headaches on a person's daily life

CONTACTS AND LOCATIONS:
Overall Officials: Xavier Moisset, Principal Investigator — CHU de Clermont-Ferrand; Cristina Alba-Delgado, Principal Investigator — Université d'Auvergne
Locations (1):
- CHU de Clermont-Ferrand, Clermont-Ferrand, France

IPD SHARING:
Plan to Share IPD: No